CLINICAL TRIAL: NCT02921399
Title: Optimal Initiation of Helicobacter Pylori Eradication After Endoscopic Resection
Brief Title: Optimal Initiation of Helicobacter Pylori Eradication After Endoscopic Resection for Gastric Neoplasm
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Hoon Youn, Department of Internal Medicine,, Gangnam Severance Hospital
Other Study IDs: 3-2016-0175
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: H.Pylori Eradication Rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early eradication group: In the post-endoscopic resection period, patients were grouped by timing (i.e., initiation) of therapy to eradicate H. pylori as follows: 1) early (≤ 2 weeks), 2) late (≥ 8weeks).
  Interventions: Other: eradication timing
- late eradication group: In the post-endoscopic resection period, patients were grouped by timing (i.e., initiation) of therapy to eradicate H. pylori as follows: 1) early (≤ 2 weeks), 2) late (≥ 8weeks).
  Interventions: Other: eradication timing

INTERVENTIONS:
Other: eradication timing — patients who underwent ESD for gastric neoplasms were randomized to receive early (3-5 days) or late (8-9 weeks) H. pylori eradication therapy after ESD.

SUMMARY:
After endoscopic resection (ER) of gastric tumors, eradication of Helicobacter pylori (H. pylori) infection is advised to reduce metachronous recurrence. However, few studies have addressed factors influencing H. pylori eradication rates in the aftermath of ER, and none have focused on the optimal timing of therapy to eradicate H. pylori post-ER.Therefore, the investigators will conduct to evaluate whether differences in timing of eradication therapy after ER of gastric tumors.

DETAILED DESCRIPTION:
Uur previous retrospective study unveiled that administering eradication treatment within 2 weeks post-ESD during the active reparative phase of ESD-induced ulcers yielded a markedly higher success rate compared to treatment post-8 weeks during the scarring phase of ESD-induced ulcers.Therefore, we conducted a multicenter, randomized, prospective study to ascertain whether the optimal timing of eradication post-ESD could influence the eradication success rate.

ELIGIBILITY:
Inclusion Criteria:

1. patients underwent endoscopic resection of gastric neoplasm
2. patients who diagnosed as H. pylori infection by rapid urease test

Exclusion Criteria:

1. Histories of gastric surgery
2. Histories of prior H. pylori eradication therapy
3. Use of drugs affecting H. pylori positivity (proton pump inhibitor, histamine-2 receptor blocker, or antibiotics) within the preceding 2 weeks

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received proton-pump inhibitor (PPI)-based triple therapy for H. pylori eradication after endoscopic resection for gastric neoplasms. Clinicopathologic characteristics, particularly the timing of triple therapy, were used to compare eradication rates, assigning patients to early- (≤2 weeks),and late-phase (≥8 weeks) eradication groups.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate according to timing of therapeutic regimen after endoscopic resection | The success of H. pylori eradication was determined using a urea breath test conducted 13 weeks ± 5 days after ESD
  The success of H. pylori eradication was determined using a urea breath test conducted

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Yonsei Unversity, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh CW, Jung DH, Kim JH, Park H, Youn YH. Early versus Late Eradication of Helicobacter pylori after Endoscopic Submucosal Dissection of Gastric Neoplasms: A Prospective, Multicenter, Randomized, Controlled Study. Gut Liver. 2025 Nov 15;19(6):821-828. doi: 10.5009/gnl250004. Epub 2025 May 28. PMID 40425226